CLINICAL TRIAL: NCT03168490
Title: In Vivo Human Intervention Approach to Test the Effects of "Gluten Friendly Bread" in Coeliac Disease Patients: GLUTEN FRIENDLY STUDY
Brief Title: In Vivo Effects of the Gluten Friendly Bread in Coeliac Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Life Sciences Department, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LSC 15/146
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: A single-centre, prospective, randomised, placebo-controlled, parallel-group trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1.5g low gluten friendly bread (Active Comparator): 1.5g low gluten friendly bread as15g bun/day to be consumed as 250 ml beverages at breakfast for 14 days
  Interventions: Dietary Supplement: Gluten Friendly bread
- 3g medium gluten friendly bread (Active Comparator): 3g medium gluten friendly bread as 30g bun to be consumed as 250 ml beverages at breakfast for 14days
  Interventions: Dietary Supplement: Gluten Friendly bread
- 6g high gluten friendly bread (Active Comparator): 6g high gluten friendly bread as 60g bun to be consumed as 250 ml beverages at breakfast for 14 days
  Interventions: Dietary Supplement: Gluten Friendly bread
- Control bread (Placebo Comparator): Placebo control bread as 15g bun to be consumed as 250 ml beverages at breakfast for 14 days
  Interventions: Dietary Supplement: Gluten Friendly bread
- Gluten free bread (Placebo Comparator): Gluten bread as 15g bun to be consumed as 250 ml beverages at breakfast for 14 days
  Interventions: Dietary Supplement: Gluten Friendly bread

INTERVENTIONS:
Dietary Supplement: Gluten Friendly bread — parallel study

SUMMARY:
In the last two decades, a series of epidemiological studies have shown a particular increase in Coeliac Disease (CD), a life-long intolerance to gluten proteins (the seed storage proteins) present in most cereals (wheat, barley and rye) both in the United States and Europe, and in developing countries. In these subjects, the consumption of cereals containing gluten causes a chronic inflammatory process leading to lesions in the small intestine and a dysfunction in nutrient absorption.The only current treatment for CD is a strict lifelong gluten-free diet. In most cases (some people do not respond) this dietary regimen guarantees the full recovery of small intestine architecture and functions, though for many patients the gluten-free diet is highly restrictive, especially for social events and during travelling. In addition, this dietary therapy has often low content of vitamins and ions, such as vitamins B and calcium, iron, zinc and magnesium, as well as fibre. Furthermore, one of the major risks is to develop obesity and diseases related to metabolic syndrome.

Recently a new and innovative detoxification method has been developed with the purpose to overcome the disadvantages of the prior methods. The method is based on the application of microwave energy for few seconds to hydrated wheat kernels; the treatment induces modifications to endosperm components which dramatically reduce the immunogenicity of the most common epitopes involved in coeliac disease, without compromising the technological properties necessary to process flour into bread, pasta and other baked goods.

The method is based on the analysis of recent studies that have reported, when high temperatures are applied to the caryopsis of wheat, the protein polymers present in the pasta produced with these "baked grain" present a size distribution pattern that is not observed in pasta during the drying cycles. The researchers Lamacchia and others explained this phenomenon on the basis of the fact that in the caryopsis of wheat, gluten is not yet formed and gluten proteins are deposited in different protein bodies.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of gluten friendly bread on the faecal microbiota composition, metabolism and immunity in coeliac individuals aged 20-80 years.

The study consists of a 6-visit (screening visit + 5 visits) randomised intervention with the Gluten Friendly bread at different doses and placebo (control bread).

Subjects will be randomly distributed into four groups: placebo (control bread in a dose of 1.5 g gluten/day), low gluten group taking the Gluten Friendly bread in a dose of 1.5 g gluten/day, medium gluten group (3 g gluten/day) and high gluten group (6 g gluten/day). As wheat generally contains 10% of gluten (i.e. 100 g of bread contain 10 g of gluten), bread buns of 60 g, 30 g and 15 g will be elaborated for high, medium and low gluten groups, respectively.

Control bread and also gluten free bread as 15g buns will be assessed as controls.

The study will include a screening visit, baseline visit, visits at midpoint, endpoint of the treatment periods and a final visit after 2 weeks of the treatment. Volunteers will provide a blood sample at a pre- screening visit (~10ml; 1 dessert spoon), to check for anaemia (defined as haemoglobin men <14g/dl; women <11.5g/dl). The design will include a 14-day run-in period followed by 14 days of treatment and a final visit post-gluten challenge. Participants will be asked to consume a multi-sugar drink (7.5g lactulose and 2g D-mannitol ≥98% in 100 ml of water) (a dosage used widely in oral clinical testing- LAMA testing) in the evening before each study visit (visits: 1, 2, 3, 4 and 5) at 8 pm and be instructed to collect all overnight and morning first spot pass urine sample. This non-invasive assessment of intestinal permeability in humans has a 20-year history. LAMA evaluation has been reported to be an accurate measure of small intestinal mucosal permeability though assessment of differential absorption of lactulose and mannitol. They will also provide a faecal sample for each study visit (visits: 1, 2, 3, 4 and 5).

Each visit will take approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20-80 years of age
* Have a medical diagnosis for coeliac disease (blood test and biopsy confirmed)
* On a gluten-free diet for a minimum of 12 months
* Able to attend 6 appointments and donate blood, urine and faecal samples before and after bread intake
* Willing to participate in the entire study (signed informed consent required)

Exclusion Criteria:

* History or evidence of intestinal disease; such as tumour, irritable bowel syndrome, etc., within the previous 5 years
* Diagnosed with another auto-immune condition (e.g. Type 1 diabetes, autoimmune thyroid disease)
* Be extremely sensitive to exposure to gluten
* Received antibiotics in the previous six months
* History of malignancy within the previous 5 years (with exception of well-treated basal cell carcinoma or in situ cervical carcinoma)
* Smoker
* Lactose intolerant
* Currently prescribed immunosuppressive drugs. Participants will be required to withdraw should they begin taking any of the ineligible medication
* Intention to use regularly other medication which affects gastrointestinal motility
* History of alcohol or drug misuse
* Suffer from any major conditions involving the following:
* Head
* Ears
* Eyes
* Nose and Throat
* Dermatological/Connective tissue
* Neurological
* Lymphatic
* Urogenital/Rectal
* Abdominal
* Respiratory
* A previous cardiovascular event within the last 6 months
* presence of secondary dyslipemias related to thyroid dysfunction
* used any drug affecting lipid metabolism in previous 3 months
* a history of alcohol abuse

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
The cellular and molecular basis for modulation of immune function by GLUTEN FRIENDLY BREAD | Change from baseline at 14 days
  Blood samples will be processed and analyzed for inflammatory/immune biomarkers (trans-glutaminase IgA and IgG, cytokines INF-Ɣ, IL-6, IL-8, IL-10, TNF-α and C-reactive protein).
  activation markers, expression of toll like receptors.

SECONDARY OUTCOMES:
The modulation of the gut microbiota by gluten friendly bread | Change from baseline at 14 days
  Fecal16S rRNA amplicon sequencing to assess changes in fecal bacterial abundance and species diversity

OTHER OUTCOMES:
Digestive symptoms | Change from baseline at 14 days
  Bristol stool scale
Microbiota activity (intestinal gas production) | Change from baseline at 14 days
  Intestinal gas evacuation on standardized diet
Intestinal gut permeability | Change from baseline at 14 days
  by measuring the urinary excretion of sugars after the ingestion of a multi-sugar drink

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Lamacchia, Study Director — The University of Foggia-Italy
Locations (1):
- Health Sciences Research Centre, Life Sciences Department, University of Roehampton, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No